CLINICAL TRIAL: NCT03421405
Title: Assessing Repeatability of NeuroCatch Platform™ Measurements: An Initial Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NCI_NCClin_001
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Brain Health

STUDY DESIGN:
Intervention Model Description: All participants will be asked to attend 4 separate experimental sessions over the course of approximately 4 weeks (i.e. one session/week). During each session, participants will listen to three different auditory stimulus sequences including sounds and words while EEG activity is recorded. There will be 5-minute break between each audio sequence. Each experimental session will take approximately 30-45 minutes to complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): All participants will be asked to attend 4 separate experimental sessions over the course of approximately 4 weeks (i.e. one session/week). During each session, participants will listen to three different auditory stimulus sequences including sounds and words while EEG activity is recorded using the NeuroCatch Platform™ device.
  Interventions: Device: NeuroCatch Platform™

INTERVENTIONS:
Device: NeuroCatch Platform™ — NeuroCatch Platform™ consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP) information.

SUMMARY:
EEG signals have been collected and studied since the early 1990's as a way of assessing brain function at a gross level. As early as the 1930's a derivative of the raw EEG signal - event-related potentials (ERPs) - have been computed. These scalp-recorded ERPs are the brains response to a stimulus of interest (e.g. a flashing checkerboard or an angry face). The timing and topographical location of ERP components lends insight into the timing and complexity of various cognitive processes. At NeuroCatch Inc., research is primarily focused on three ERP components: the N100, P300 and N400.

To elicit the ERP components of interest in this study (N100, P300, N400), proprietary auditory stimulus sequences will be administered using the investigational device, the NeuroCatch Platform™. Each sequence consists of pure tones and word pairs to elicit the various components associated with different attention abilities (sensory processing, target detection & semantic processing). A secondary objective of the study will be to validate the auditory stimulus sequences tested.

Understanding the degree to which these neurophysiological components fluctuate over time is crucial to our understanding of typical brain functioning. Research and medicine is moving away from behavioural responses to assess brain health (e.g. verbal responses, reaction time, etc.) and are moving toward more neuroimaging focused measures, such as CT, and MRI scans. The strength of utilizing EEG technology is two-fold: i) it is portable and ii) has high temporal resolution. Looking forward, EEG-based brain assessment technology could be implemented field-side, at the site of an accident for a quick assessment of brain and cognitive functioning, or within a clinicians' office to evaluate treatment efficacy. However, for this type of technology to be useful in quantifying brain health, we must first quantify the degree to which a healthy brain naturally fluctuates in it processing capability. For example, should technology such as the NeuroCatch Platform™ be used as a monitoring tool, we must have an idea of what normal variation is.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 19-65 years old inclusively
2. Normal hearing capabilities
3. Able to understand the informed consent form, study procedures and willing to participate in study
4. Able to keep eyes still for min 6 minutes

Exclusion Criteria:

1. Clinically documented hearing issues (e.g. tinnitus, in-ear hearing problems, punctured ear drum, etc.)
2. Implanted pacemaker
3. Metal or plastic implants in skull
4. In-ear hearing aid or chocclear implant, hearing device
5. Chronic neurological disorder (e.g. Stroke, MS, etc.)
6. Recent (within last 6 months) acquired brain injury
7. History of brain cancer
8. History of dementia
9. Exposed to investigational drug or device 30 days prior to start in this study, or concurrent use of investigational drug or device while enrolled in this study
10. Planning to use investigational drugs or devices while enrolled in this study
11. Not fluent in English language
12. Unable to provide informed consent
13. Previous participation in studies using the NeuroCatch Platform™
14. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
15. History of seizures
16. Allergy to rubbing alcohol or EEG gel

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Variability of response size of selected ERPs (N100, P300, N400) acquired using the NeuroCatch Platform™ during the baseline visit | 1 day
  Response size will be measured as amplitude in microvolts.
Variability of response timing of selected ERPs (N100, P300, N400) acquired using the NeuroCatch Platform™ during the baseline visit | 1 day
  Response timing will be measured as latency in milliseconds.

SECONDARY OUTCOMES:
Qualitative comparison of ERP graphs generated by different auditory stimulus sequences during the NeuroCatch Platform™ assessment | 1 day
  ERP graphs will be overlaid. Trained technician will assess if peaks and valleys occur at expected time points for different sequences.
Collection and evaluation of adverse events and adverse device effects | 4 weeks
  Evaluation of safety and tolerability of the NeuroCatch Platform™ device
Slope of change over time in response size to quantify the natural variability in selected ERPs (N100, P300, N400) acquired using NeuroCatch Platform™ | 4 weeks
  Response size will be measured as amplitude in microvolts. Means will be calculated and compared over time.
Slope of change over time in response timing to quantify the natural variability in selected ERPs (N100, P300, N400) acquired using NeuroCatch Platform™ | 4 weeks
  Response timing will be measured as latency in milliseconds. Means will be calculated and compared over time.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Venter, MBChB MFamMed CCFP IFMCP, Principal Investigator — HealthTech Connex Inc. Centre for Neurology Studies
Locations (1):
- HealthTech Connex Inc. Centre for Neurology Studies, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided